CLINICAL TRIAL: NCT02055066
Title: A Phase 1b Study of ARGX-111 in Patients With Advanced Cancer Over-expressing the c-Met Protein.
Brief Title: A Phase 1b Study of ARGX-111 in Patients With Advanced Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-111-1301
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: cancer; c-MET
MeSH Terms: conditions — Neoplasms | interventions — ARGX-111

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): ARGX-111 0.3 mg/kg
  Interventions: Drug: ARGX-111
- Arm 2 (Experimental): ARGX-111 1.0 mg/kg
  Interventions: Drug: ARGX-111
- Arm 3 (Experimental): ARGX-111 3.0 mg/kg
  Interventions: Drug: ARGX-111
- Arm 4 (Experimental): ARGX-111 10 mg/kg
  Interventions: Drug: ARGX-111

INTERVENTIONS:
Drug: ARGX-111

SUMMARY:
This a first-in-human study of an antibody blocking the function of the oncogene c-met in patients with cancer.

DETAILED DESCRIPTION:
This Phase 1b trial will characterize the safety profile of ARGX 111 and will thus provide the first elements towards establishing an accurate risk-benefit assessment for ARGX 111 in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age ≥ 18 years.
3. Performance status of 0 or 1.
4. Histological diagnosis of malignancy.
5. Cancer relapsing after, or refractory to standard therapy.
6. Malignancy over-expressing the c Met protein.
7. Presence of circulating tumor cells (CTCs).
8. At least one tumor lesion > 2 cm on PET/CT.
9. Serum albumin > 35 g/L.
10. Absolute neutrophil count (ANC) > 1.0 x 109/L.
11. Hemoglobin > 90 g/L (0.9 g/dL).
12. Platelet count ≥ 75 x 109/L.
13. Coagulation parameters ≤ 1.5 x ULN.
14. Total bilirubin ≤ 1.5 x upper limit of normal (ULN).
15. Creatine Phosphokinase (CPK) ≤ 2.5 x ULN.
16. Serum creatinine ≤ 1.5 x ULN.
17. Ability to comply with protocol-specified procedures/evaluations and scheduled visits.

Exclusion Criteria:

1. History or clinical evidence of neoplastic central nervous system (CNS) involvement.
2. Major surgery within 4 weeks of ARGX 111 first dose administration.
3. Systemic glucocorticoid administration at doses greater than physiological replacement (prednisone 20 mg equivalent) within 3 weeks of ARGX 111 first dose administration.
4. Cytotoxic chemotherapy within 3 weeks of ARGX 111 first dose administration.
5. Radiation therapy with curative intent within 3 weeks of ARGX 111 first dose administration.
6. Biological therapy (monoclonal antibodies) within 4 weeks of ARGX 111 first dose administration.
7. Biological therapy (other than monoclonal antibodies) within 5 half-lives of ARGX 111 first dose administration.
8. Unresolved Grade 3 or 4 toxicity from prior therapy, including experimental therapy.
9. History of recurrent Grade 3 or 4 toxicity from anti c Met therapy.
10. Uncontrolled diabetes, defined as fasting glycemia > 150 mg/dl).
11. Active, untreated viral, bacterial, or systemic fungal infection.
12. Any clinical finding, including psychiatric and behavioral problems, which, in the opinion of the Investigator, precludes the patient from safely participating in the study.
13. Childbearing potential (unless using an adequate measure of contraception).
14. Pregnancy or lactation.
15. History of severe (Grade 3 or 4) hypersensitivity to recombinant proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 1 month
  Number of patients with grade 3 or 4 toxicity

SECONDARY OUTCOMES:
Pharmacokinetic profiles (Cmax , Ctrough, AUC, Vd , clearance, and half-life) | C1 D1 (pre, 0h, 2h, 6h, 12h, 24h), C1D8, C1D15; Cycle ≥2 o D1 pre-/post-dose
  Measurement of drug concentration in the blood
Biomarkers (Hepatocyte growth factor; ADCC) | Base-line and pre-dose at each cycle for an average of 4 months
  measurements of cytokine changes in blood as a result of drug administration
Incidence of adverse events per dose level | for an average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Awada, MD, Principal Investigator — Jules Bordet Institute
Locations (2):
- Belgium (2):
  - Universitair Zieckenhuis Antwerpen, Antwerp
  - Institut Jules Bordet, Brussels